CLINICAL TRIAL: NCT06930534
Title: Portable Rapid Imaging for Medical Emergencies
Acronym: PRIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Hyperfine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2000039013
Record Dates: First submitted 2025-03-19; First posted 2025-04-16 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Patient Satisfaction; Conventional Magnetic Resonance Imaging; Portable Magnetic Resonance Imaging
Keywords: Brain MRI
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Portable Brain MRI scan (Experimental): Participants in the scan arm will receive a portable MRI scan as soon as the scanner is available after randomization as part of their initial evaluation. Regardless of randomization arm, all participants will receive their scheduled conventional MRI as usual.
  Interventions: Device: Swoop Plus Mk2.0
- Standard of Care (No Intervention): Participants in the SOC arm will not receive a portable MRI scan as part of their initial evaluation. Regardless of randomization arm, all participants will receive their scheduled conventional MRI as usual.

INTERVENTIONS:
Device: Swoop Plus Mk2.0 — portable brain MRI scanner
  Arms: Portable Brain MRI scan

SUMMARY:
This study will compare the time it takes to scan a patient in the emergency department with a portable MRI when compared to a conventional MRI. Participants will be randomized to receive a portable MRI plus standard of care (SOC) vs SOC. Investigators will look at time to beginning of scan for both.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether portable brain MRI reduces the time from scan order to scan start in the emergency department as compared to conventional brain MRI. The secondary objectives of this study are 1) to measure the percentage of scans that are completed after order and the time from order to completion, 2) to compare findings on portable MRI to conventional brain imaging findings, 3) to compare the total length of stay between the portable MRI and conventional MRI groups, and 4) to understand the impact of portable MRI scans on decision making and provider satisfaction based on qualitative surveys administered to a physician endpoint panel. This is a prospective, observational, randomized study. Participants will be recruited from the pool of patients ordered for a brain MRI, with or without contrast and excluding hyperacute MRI, in the emergency department. Participants will be randomized to one of two treatment groups, scan or standard-of-care (SOC). Participants in the scan arm will receive a portable MRI scan as soon as the scanner is available after randomization.

Participants in the SOC arm will not receive a portable MRI scan as part of their initial evaluation. Regardless of randomization arm, all participants will receive their scheduled conventional MRI as usual. Information on each participant's clinical course, conventional imaging, and length of stay will be collected, regardless of treatment group. On a rolling basis, surveys containing deidentified clinical information and portable MRI scans will be administered to a physician panel to assess the impact of portable MRI scans on decision making and provider satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age at presentation to Yale New Haven Hospital Adult ED
* Order to receive conventional brain MRI imaging originating in the YNHH Adult ED

Exclusion Criteria:

* Lack of assent from treating physician for inclusion in this protocol.
* Contraindications to 1.5T MRI evaluation, including:

  1. Cardiac Pacemaker or defibrillator
  2. Aneurysm clip
  3. Implants or devices attached to the body in the chest or above, such as:

     1. Nerve stimulator
     2. Deep brain stimulator
     3. Programmable shunt
     4. Stent
     5. Pain pump
     6. Artificial extremity
  4. Implants in the ears (hearing aid or cochlear implant
  5. Any shrapnel, pellets, bullets, metallic fragments, or other metallic foreign body above the chest
  6. Metallic joints, rods, screws, or other orthopedic implants in or above the chest
  7. Braces, dentures, removable teeth, or dental expanders that cannot be removed.
  8. Body piercings in or above the chest that cannot be removed.
  9. MRI-incompatible Tracheostomy tube or Swan Ganz catheter in place
  10. Status Epilepticus or anyone previously seizing deemed by the physician not to be suitable for pMRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Time to start of scan | immediately post MRI (Day 1)
  Time from brain MRI order to start of scan, either portable or conventional.

SECONDARY OUTCOMES:
Percentage of Completed Scans | immediately post MRI (Day 1)
  The proportion of scans completed in each arm will be compared.
Portable MRI Findings | immediately post MRI (Day 1)
  The frequency of acute findings (e.g., ischemic stroke, intracranial hemorrhage) using the portable MRI will be compared between groups.
Length of Stay | immediately post MRI (Day 1)
  Total Emergency Department length of stay
Provider Satisfaction Survey | immediately post MRI (Day 1)
  Provider survey data will be summarized using descriptive statistics and thematic analysis for qualitative responses.
Non-Completed Scans | immediately post missed MRI (Day 1)
  To document the reasons for non-completion of MRI scans

CONTACTS AND LOCATIONS:
Overall Officials: Adam de Havenon, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Health Emergency Department, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No